CLINICAL TRIAL: NCT05482945
Title: CardioPulmonary Resuscitation With Argon (CPAr) Trial
Acronym: CPAr
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRFMN-7557
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Cardiac Arrest With Successful Resuscitation
Keywords: Cardiac arrest; Cardiopulmonary resuscitation; Argon.
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Intervention Model Description: The intervention (Ar/O2 or standard ventilation) is assigned to the patient using a centrally generated randomization plan, balanced by centre.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients will be ventilated with a mixture of Ar 70%/O2 30% for 4 hours
  Interventions: Drug: Noble gas Argon
- Control-standard (No Intervention): Ventilation with a FiO2 of 30% in room air is continued for 4 hours.

INTERVENTIONS:
Drug: Noble gas Argon — Ventilation with Ar 70%/O2 30% in comatose patients resuscitated from OHCA with the use of an experimental mechanical ventilator.
  Arms: Intervention

SUMMARY:
Preclinical studies suggest that argon (Ar) might diminish the neurological and myocardial damage after any hypoxic-ischemic insult. Indeed, Ar has been tested in different models of ischemic insult, at concentrations ranging from 20% up to 80%. Overall, Ar emerged as a protective agent on cells, tissues and organs, showing less cell death, reduced infarct size and faster functional recovery. More specifically, encouraging data has been reported in animal studies on cardiac arrest (CA) in which a better and faster neurological recovery was achieved when Ar was used in the post-resuscitation ventilation. More importantly, these benefits have been replicated in different studies, enrolling both small and large animals. Finally, ventilation with Ar in O2 has been demonstrated to be safe both in animals and humans. Based on this evidence, a clinical translation is advocated. Thus, the CardioPulmonary resuscitation with Argon - CPAr trial has been conceived. The trial initially started as phase I-II trial to specifically address the question about the safety of the post resuscitation Ar-treatment. The available data on the first 30 randomized patients, evaluated by the Data Safety Monitoring Board (DSMB), were considered absolutely reassuring with regard to the safety of the experimental treatment. In this perspective, the DSMB supported the continuation of the study as a phase II trial, maintaining the study protocol in all its aspects. Thus, the aim of the CPAr trial is now to evaluate efficacy in reducing post-CA neurological injury of Ar/O2 ventilation in patients resuscitated from CA.

DETAILED DESCRIPTION:
The trial is a multicenter, randomized, controlled, single blinded, phase II and pre marketing study in patients resuscitated from Out-of-hospital cardiac arrest (OHCA).

All eligible patients will be treated in full and documented compliance with the European ResuscitationCouncil (ERC)/European Society of Intensive Care Medicine (international guidelines and local post resuscitation protocols). In addition, a randomized assignment ensures a strict comparability for both the periods of data collection of safety end-points (to be assessed blindly by the events Committee): the four hours of duration of study treatment, and the longer period of possibly related clinical events during 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission after resuscitation from witnessed non-traumatic out-of-hospital cardiac arrest (OHCA) of presumably cardiac etiology with a presenting shockable rhythm;
* age ≥ 18 years;
* unconsciousness after return of spontaneous circulation (ROSC);
* duration of CPR ≤ 40 mins;
* initiation of study intervention ≤ 4 hrs from ROSC;
* stable SaO2 ≥ 94% with a FiO2 of 30%.

Exclusion Criteria:

* Non-witnessed CA;
* CA of traumatic origin or from a non-presumably cardiac cause;
* CA with a non-shockable presenting rhythm (pulseless electrical activity and asystole);
* female of childbearing potential defined as younger of 50 years;
* pregnancy;
* known terminal illness;
* pre-CA cerebral performance category (CPC) ≥ 3;
* initiation of the study intervention > 4 hrs from ROSC;
* participation to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Neuronal preservation | 48 hours
  Efficacy of Argon treatment in reducing post-CA neurological injury, assessed as 48hr serum concentration of the Neuron Specific Enolase (NSE), an established biomarker of brain injury.

SECONDARY OUTCOMES:
Myocardial preservation | Up to 96 hours
  Ar effect on myocardial protection is assessed through measure of hs-cTnT release
Brain injury | 96 hours
  Ar effect on brain injury is assessed through MRI (imaging) if patient remains comatose
Survival | ICU discharge (assessed up to 7 days), 1-month, 6 months
  Effect of argon on survival after cardiac arrest (days)
Neurological recovery | ICU discharge (assessed up to 7 days), 1-month, 6 months
  Neurological functional recovery is assessed with the CPC score
Multiorgan function | Up to 96 hours
  Multiorgan function is assessed through the evaluation of sequential organ failure assessment score (SOFA). The score sequentially assesses the presence and severity of dysfunctions in six organ systems: respiratory, cardiovascular, coagulation, hepatic, neurological and renal scoring 0 to 4 points per each one of the following:
  PaO2-fiO2 ratio; Mean arterial pressure (mmHg) or vasoactive treatment; Creatinine (mg/dL) or 24-h diuresis (ml/24h); Platelet count (x103/mm3); Serum bilirubin (mg/dL); Glasgow coma scale
  The following markers are also assessed:
  transaminases (UI/L) Pancreatic amilase, lipase (UI/L)
Incidence of Treatment-Emergent Adverse Events | 1 month
  The incidence, the timing, and the duration of the need to stop Ar 70% treatment in order to maintain the SPO2> 90%.
  The incidence of potentially Ar-attributable hemodynamic adverse events (i.e. arterial hypotension not responsive to fluids and/or vasoactive/inotropic drugs).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Ristagno, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (9):
- Italy (9):
  - Ospedale Policlinico San Martino di Genova, Genova, GE
  - Ospedale San Gerado, Monza, MB
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan
  - Azienda Ospedaliero - Universitaria di Parma, Parma, Parma
  - Ospedale Civile Santa Maria degli Angeli di Pordenone, Pordenone, Pordenone
  - Arcispedale Santa Maria Nuova di Reggio Emilia, Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Ospedale Santa Chiara di Trento, Trento, Trento
  - Azienda Sanitaria Universitaria Giuliano Isontina (Asugi) di Trieste, Trieste, TS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ristagno G, Staszewsky L, Merigo G, Magliocca A, Cucino A, Meessen J, Fumagalli F, Pozzi M, Galazzi A, Sandroni C, Meneguzzi M, Marangone A, Robba C, Roman-Pognuz E, Salati G, Picetti E, Novelli D, Bellani G, Panigada M, Wik L, Garattini S, Foti G, Antonelli M, Zanier E, Grasselli G, Latini R; CPAr Study group. CardioPulmonary resuscitation with Argon (CPAr): A protocol for a randomised controlled multicentre clinical trial. Resusc Plus. 2025 Sep 10;26:101096. doi: 10.1016/j.resplu.2025.101096. eCollection 2025 Nov. PMID 41079544